CLINICAL TRIAL: NCT00718952
Title: Multi-centre, Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Treatment of Pulmonary Arterial Hypertension With Vardenafil in China
Brief Title: The Efficacy and Safety of Vardenafil in the Treatment of Pulmonary Arterial Hypertension
Acronym: EVALUATION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Professor Zhi-Cheng JING, Shanghai Pulmonary Hospital, Tongji University,Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVALUATION-01
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients in group A will receive vardenafil in double-blinded treatment period.
  Interventions: Drug: Vardenafil
- B (Placebo Comparator): Patients in group A will receive placebo in double-blinded treatment period.
  Interventions: Drug: Placebo; Drug: Vardenafil

INTERVENTIONS:
Drug: Vardenafil — vardenafil tablet 5mg once-daily orally in the first 4 weeks while 5mg twice-daily orally in the following 8 weeks.
  Other Names: Levitra
  Arms: A
Drug: Placebo — Placebo tablet 5mg once-daily orally in the first 4 weeks while 5mg twice-daily orally in the following 8 weeks.
  Arms: B
Drug: Vardenafil — Patients in all the 2 arms will take vardenafil tablet 5mg twice-daily orally from week 13 to week 24(open-label).
  Other Names: Levitra

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vardenafil in the treatment of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), defined as a mean pulmonary artery pressure ≥25 mmHg with a pulmonary capillary wedge pressure ≤15 mmHg measured by cardiac catheterization, is a disorder that may occur either in the setting of a variety of underlying medical conditions or as a disease that uniquely affects the pulmonary circulation. Irrespective of its etiologies, PAH is a serious and often progressive disorder that results in right ventricular dysfunction and impairment in activity tolerance, and may lead to right-heart failure and death. The pathogenesis of PAH is complex and incompletely understood, but includes both genetic and environmental factors that alter vascular structure and function.

In recent years, several new drugs have been developed for the treatment of pulmonary arterial hypertension (PAH), including continuous intravenous epoprostenol, inhaled iloprost, subcutaneous trepostinil, oral bosentan, and oral beraprost. In addition, there is increasing evidence for the therapeutic effectiveness of the phosphodiesterase-5 (PDE-5) inhibitor sildenafil in PAH. Phosphodiesterases are a superfamily of enzymes that inactivate cyclic adenosine monophosphate and cyclic guanosine monophosphate, the second messengers of prostacyclin and nitric oxide (NO) .The phosphodiesterases have different tissue distributions and substrate affinities. Interestingly, PDE-5 is abundantly expressed in lung tissue, thus offering as target molecule for PAH treatment concepts.

The three commercially available PDE-5 inhibitors (sildenafil, vardenafil, and tadalafil) are currently approved for the treatment of erectile dysfunction . These inhibitors are now receiving attention for their activity in the pulmonary vasculature. Sildenafil has been proved to improve the exercise capacity and pulmonary hemodynamics of PAH patients, however, there are few reports regarding the use of vardenafil or tadalafil on the pulmonary vasculature. Although sildenafil, vardenafil, and tadalafil act on the same enzyme, these drugs exhibit different pharmacokinetics and selectivity, and therefore may not be equally efficacious in the pulmonary vascular bed. As vardenafil has a more than 20-fold greater potency than sildenafil for inhibiting purified PDE-5, we assume that it will show more favorable clinical and side-effect profiles in treating PAH.

This is a prospective, randomized, placebo-controlled, pilot study to evaluate the efficacy and safety of vardenafil in the treatment of pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 12-65.
* Confirmed idiopathic pulmonary hypertension, connective tissue disease associated pulmonary hypertension, congenital heart disease(with Eisenmenger syndrome) associated pulmonary hypertension.
* Baseline 6-minutes walking distance 150m-550m.
* WHO pulmonary hypertension function II-III with non-responder to calcium channel blockers.
* Documented written informed consent.

Exclusion Criteria:

* The other types of pulmonary hypertension.
* Subjects who refuse to subscribe written informed consents or can't cooperate with the trial well.
* Subjects with serious acute or chronic disease involved liver, kidney, and brain or have to use potent CYP3A4-inhibitor or nitrate to treat the underlying diseases.
* Subjects who are currently treated with sildenafil for PAH or taking sildenafil or tadalafil.
* Other contraindications in package insert.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The change in exercise capacity, as measured by the total distance walked in six minutes | at week 12 and week 24

SECONDARY OUTCOMES:
The reduction of mean pulmonary-artery pressure(mPAP)and pulmonary vascular resistance(PVR) | at week 12 and week 24
The increase of cardiac output(CO) | at week 12 and week 24
The increase of Peripheral Saturation of oxygen(SPO2) | at week 12 and week 24
The change in the Borg dyspnea index(a measure of perceived breathlessness on a scale of 0 to 10, with higher values indicating more severe dyspnea) | at week 12 and week 24
The change in World Health Organization (WHO) functional classification of pulmonary arterial hypertension (an adaptation of the New York Heart Association classification) | at week 12 and week 24
Time from randomization to clinical worsening(defined as death, transplantation,hospitalization for PAH and worse right heart failure,acute heart failure,or vardenafil allergy,or worsening leading to discontinuation,need for epoprostenol or bosentan) | From baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Cheng Jing, MD, Principal Investigator — Shanghai Pulmonary Hospital Affiliated to Tongji University, Shanghai, China
Locations (9):
- China (9):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Hospital, Peking Union Medical College, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Peking University, Beijing, Beijing Municipality
  - The First Clinical College of Harbin Medical University, Harbin, Heilongjiang
  - Xiangya Hospital, Central-South University, Changsha, Hunan
  - The General Hospital of Shenyang Military Command, Shenyang, Liaoning
  - Renji Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Medical College of Xian Jiaotong University, Xi’an, Shanxi
  - Shanghai Pulmonary Hospital ,Tongji University, Shanghai

REFERENCES:
- [Background] Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, Groves BM, Tapson VF, Bourge RC, Brundage BH, Koerner SK, Langleben D, Keller CA, Murali S, Uretsky BF, Clayton LM, Jobsis MM, Blackburn SD, Shortino D, Crow JW; Primary Pulmonary Hypertension Study Group. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1996 Feb 1;334(5):296-301. doi: 10.1056/NEJM199602013340504. PMID 8532025
- [Background] Olschewski H, Simonneau G, Galie N, Higenbottam T, Naeije R, Rubin LJ, Nikkho S, Speich R, Hoeper MM, Behr J, Winkler J, Sitbon O, Popov W, Ghofrani HA, Manes A, Kiely DG, Ewert R, Meyer A, Corris PA, Delcroix M, Gomez-Sanchez M, Siedentop H, Seeger W; Aerosolized Iloprost Randomized Study Group. Inhaled iloprost for severe pulmonary hypertension. N Engl J Med. 2002 Aug 1;347(5):322-9. doi: 10.1056/NEJMoa020204. PMID 12151469
- [Background] Simonneau G, Barst RJ, Galie N, Naeije R, Rich S, Bourge RC, Keogh A, Oudiz R, Frost A, Blackburn SD, Crow JW, Rubin LJ; Treprostinil Study Group. Continuous subcutaneous infusion of treprostinil, a prostacyclin analogue, in patients with pulmonary arterial hypertension: a double-blind, randomized, placebo-controlled trial. Am J Respir Crit Care Med. 2002 Mar 15;165(6):800-4. doi: 10.1164/ajrccm.165.6.2106079. PMID 11897647
- [Background] Rubin LJ, Badesch DB, Barst RJ, Galie N, Black CM, Keogh A, Pulido T, Frost A, Roux S, Leconte I, Landzberg M, Simonneau G. Bosentan therapy for pulmonary arterial hypertension. N Engl J Med. 2002 Mar 21;346(12):896-903. doi: 10.1056/NEJMoa012212. PMID 11907289
- [Background] Galie N, Humbert M, Vachiery JL, Vizza CD, Kneussl M, Manes A, Sitbon O, Torbicki A, Delcroix M, Naeije R, Hoeper M, Chaouat A, Morand S, Besse B, Simonneau G; Arterial Pulmonary Hypertension and Beraprost European (ALPHABET) Study Group. Effects of beraprost sodium, an oral prostacyclin analogue, in patients with pulmonary arterial hypertension: a randomized, double-blind, placebo-controlled trial. J Am Coll Cardiol. 2002 May 1;39(9):1496-502. doi: 10.1016/s0735-1097(02)01786-2. PMID 11985913
- [Background] Ghofrani HA, Wiedemann R, Rose F, Olschewski H, Schermuly RT, Weissmann N, Seeger W, Grimminger F. Combination therapy with oral sildenafil and inhaled iloprost for severe pulmonary hypertension. Ann Intern Med. 2002 Apr 2;136(7):515-22. doi: 10.7326/0003-4819-136-7-200204020-00008. PMID 11926786
- [Background] Michelakis E, Tymchak W, Lien D, Webster L, Hashimoto K, Archer S. Oral sildenafil is an effective and specific pulmonary vasodilator in patients with pulmonary arterial hypertension: comparison with inhaled nitric oxide. Circulation. 2002 May 21;105(20):2398-403. doi: 10.1161/01.cir.0000016641.12984.dc. PMID 12021227
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] Ghofrani HA, Voswinckel R, Reichenberger F, Olschewski H, Haredza P, Karadas B, Schermuly RT, Weissmann N, Seeger W, Grimminger F. Differences in hemodynamic and oxygenation responses to three different phosphodiesterase-5 inhibitors in patients with pulmonary arterial hypertension: a randomized prospective study. J Am Coll Cardiol. 2004 Oct 6;44(7):1488-96. doi: 10.1016/j.jacc.2004.06.060. PMID 15464333